CLINICAL TRIAL: NCT04946708
Title: Using Technology to Engage Patients With Interstitial Lung Disease (ILD) in a Home a Home Exercise Program.
Brief Title: Virtual Exercise Program in Interstitial Lung Disease (ILD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Diana C Sanchez-Ramirez, PhD, Assistant professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS24936 (B2021:051)
Record Dates: First submitted 2021-06-15; First posted 2021-07-01 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Two groups pre-post assessment (pilot/feasibility study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small group zoom meeting (Experimental): Group one: will be asked to follow the exercise program with a small group of peers (2 groups/6 participants each) in a zoom meeting 3 times a week/45 min each (including 5 min before and 10 min after the meeting for free talk-chat between the participants e.g. questions, perceptions, etc.).
  Interventions: Other: Exercise program (virtual/remote)
- YouTube pre-recorded video (Experimental): Group two: will be asked to follow the exercise program 3 times a week/30 min each while watching a pre-recorded YouTube video.
  Interventions: Other: Exercise program (virtual/remote)

INTERVENTIONS:
Other: Exercise program (virtual/remote) — Intervention (8 weeks): using the participants' initial assessment and personal characteristics, the therapist will provide personalized recommendations (e.g. maximum heart rate, minimum SpO2), explain the educational materials, and instruct patients on safety precautions. All participants (and immediate caregiver if necessary) will receive training in: 1) basic device management (join a zoom meeting, watch a YouTube video), 2) use of the portable spirometer and its associated app, 3) use of finger pulse oximeter and 4) recording of the values in a dairy.

SUMMARY:
Design: this pilot-study uses a two-group random assignment pretest-posttest design. Once the groups are being selected an envelope will be mailed to the participant with the printed version of the exercise program and surveys, a portable SpiroBank Smart FN multi parameter spirometer (MIR), a finger pulse oximeter (LOOKEE), a diary, and a prepaid envelop for a subsequent post-intervention return of the equipment and surveys and the diary.

Intervention: A) Exercise program: evidence-based and user friendly educational materials with recommendations on breathing and physical exercises will be developed. B) Patients intake: in a zoom meeting, a registered therapist (Pl) in charge of implementing the intervention will request informed consent to participate in the study, explain specifics of the intervention to each participant, and will conduct an initial assessment. C) Intervention (8 weeks): using the participants' initial assessment and personal characteristics, the therapist will provide personalized recommendations (e.g. maximum heart rate, minimum Sp02), explain the educational materials, and instruct patients on safety precautions (how to pace themselves, when to seek professional or emergency care). All participants (and immediate caregiver I necessary) will receive training: 1) basic device management (join a zoom meeting, watch a YouTube video), 2) use of the portable spirometer and its associated app, 3) use of finger pulse oximeter and 4) recording of the values in a dairy. Group one: will be asked to follow the exercise program with a small group of peers (2 groups/6 participants each) in a zoom meeting 3 times a week/45 min each {including 5 min before and 10 min after the meeting for free talk-chat between the participants e.g. questions, perceptions, etc.). The therapist will lead the first three meetings, gradually encourage participants to take turns leading the exercises with the goal of identifying /empowering potential patient leaders. Beginning with the fourth meeting, participants will be encouraged to connect to the meeting and follow their exercise program on their own, taking into account their individualized recommendations. The RA will organize and attend the zoom meetings to resolve general questions (e.g. equipment, platforms, etc.) and will act as a direct point of contact between the therapist and the participants. Group two: will be asked to follow the exercise program 3 times a week/30 min each while watching a pre-recorded YouTube video. D) Self-monitoring: patients will be asked to wear the finger pulse oximeter at all times while exercising, so that they can control their pace while avoiding exceeding target values (HR, Sp02). They will be asked to record in their HR and Sp02 values before and after participation in every session of the exercise program in a diary. E) Support: participants will be able to contact the therapist at any time during the study if they have questions or concerns. Otherwise, they will receive a follow-up phone call once a week from the RA.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of interstitial lung disease
* Access to a smart phone or tablet and home internet

Exclusion Criteria:

* Acute exacerbation of their ILDs condition
* History of neurological disease or mental illness
* Inability to ambulate independently without supervision
* Inability to complete basic tasks on a smart phone or tablet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Change in lung capacity | 8 weeks
  It will be assessed using a SpiroBank Smart F/V multi parameter spirometer (MIR) at pre-post intervention and once a week in between to monitor changes. This portable spirometer, which is MDSAP approved and complaint with ATS/ERS guidelines, connects automatically via Bluetooth to an iOS & Android compatible App (MIR Spirobank). It provides real time feedback through messages and animation on smartphone, to improve personal compliance during the test. The app can generate test results PDF printout with information regarding 19 parameters of lung capacity.
Change in dyspnea | 8 weeks
  Modified Borg Scale (0 "none" to 10 "maximum") will be used to assess dyspnea.
Change in fatigue | 8 weeks
  Fatigue severity scale (0 -7 "higher worse") will be used to measure the severity of fatigue.
Change in exercise capacity | 8 weeks
  Assessed with the one-minute sit-to-stand test (number of times the persons can complete the task in one minute).
Change in post-exercise saturation | 8 weeks
  SpO2 will be measured using a digital fingertip pulse oximeter before-after the one- minute sit-to-stand test.
Change in physical function | 8 weeks
  Assessed using the EQ-5D-5L scale (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) (0-100 higher better function).
Changes in health-related quality of life (HRQoL) | 8 weeks
  Assessed with the King's Brief Interstitial Lung Disease (KBILD), which is an ILD-specific measure of HRQoL. Total score ranges are 0-100 (100 represents best HRQoL).

CONTACTS AND LOCATIONS:
Locations (1):
- U of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Travis WD, Costabel U, Hansell DM, King TE Jr, Lynch DA, Nicholson AG, Ryerson CJ, Ryu JH, Selman M, Wells AU, Behr J, Bouros D, Brown KK, Colby TV, Collard HR, Cordeiro CR, Cottin V, Crestani B, Drent M, Dudden RF, Egan J, Flaherty K, Hogaboam C, Inoue Y, Johkoh T, Kim DS, Kitaichi M, Loyd J, Martinez FJ, Myers J, Protzko S, Raghu G, Richeldi L, Sverzellati N, Swigris J, Valeyre D; ATS/ERS Committee on Idiopathic Interstitial Pneumonias. An official American Thoracic Society/European Respiratory Society statement: Update of the international multidisciplinary classification of the idiopathic interstitial pneumonias. Am J Respir Crit Care Med. 2013 Sep 15;188(6):733-48. doi: 10.1164/rccm.201308-1483ST. PMID 24032382
- [Background] Ryerson CJ, Tan B, Fell CD, Manganas H, Shapera S, Mittoo S, Sadatsafavi M, To T, Gershon A, Fisher JH, Johannson KA, Hambly N, Khalil N, Marras TK, Morisset J, Wilcox PG, Halayko AJ, Khan MA, Kolb M. The Canadian Registry for Pulmonary Fibrosis: Design and Rationale of a National Pulmonary Fibrosis Registry. Can Respir J. 2016;2016:3562923. doi: 10.1155/2016/3562923. Epub 2016 Apr 5. PMID 27445528
- [Background] Hopkins RB, Burke N, Fell C, Dion G, Kolb M. Epidemiology and survival of idiopathic pulmonary fibrosis from national data in Canada. Eur Respir J. 2016 Jul;48(1):187-95. doi: 10.1183/13993003.01504-2015. Epub 2016 May 26. PMID 27230442
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Florian J, Watte G, Teixeira PJZ, Altmayer S, Schio SM, Sanchez LB, Nascimento DZ, Camargo SM, Perin FA, Camargo JJ, Felicetti JC, Moreira JDS. Pulmonary rehabilitation improves survival in patients with idiopathic pulmonary fibrosis undergoing lung transplantation. Sci Rep. 2019 Jun 27;9(1):9347. doi: 10.1038/s41598-019-45828-2. PMID 31249363
- [Background] Dowman L, Hill CJ, Holland AE. Pulmonary rehabilitation for interstitial lung disease. Cochrane Database Syst Rev. 2014 Oct 6;(10):CD006322. doi: 10.1002/14651858.CD006322.pub3. PMID 25284270
- [Background] Dowman LM, McDonald CF, Hill CJ, Lee AL, Barker K, Boote C, Glaspole I, Goh NSL, Southcott AM, Burge AT, Gillies R, Martin A, Holland AE. The evidence of benefits of exercise training in interstitial lung disease: a randomised controlled trial. Thorax. 2017 Jul;72(7):610-619. doi: 10.1136/thoraxjnl-2016-208638. Epub 2017 Feb 17. PMID 28213592
- [Background] Hanada M, Kasawara KT, Mathur S, Rozenberg D, Kozu R, Hassan SA, Reid WD. Aerobic and breathing exercises improve dyspnea, exercise capacity and quality of life in idiopathic pulmonary fibrosis patients: systematic review and meta-analysis. J Thorac Dis. 2020 Mar;12(3):1041-1055. doi: 10.21037/jtd.2019.12.27. PMID 32274173
- [Background] Keating A, Lee A, Holland AE. What prevents people with chronic obstructive pulmonary disease from attending pulmonary rehabilitation? A systematic review. Chron Respir Dis. 2011;8(2):89-99. doi: 10.1177/1479972310393756. PMID 21596892
- [Background] Nici L, Singh SJ, Holland AE, ZuWallack RL. Opportunities and Challenges in Expanding Pulmonary Rehabilitation into the Home and Community. Am J Respir Crit Care Med. 2019 Oct 1;200(7):822-827. doi: 10.1164/rccm.201903-0548PP. No abstract available. PMID 31051091
- [Background] Spitzer KA, Stefan MS, Priya A, Pack QR, Pekow PS, Lagu T, Pinto-Plata VM, ZuWallack RL, Lindenauer PK. Participation in Pulmonary Rehabilitation after Hospitalization for Chronic Obstructive Pulmonary Disease among Medicare Beneficiaries. Ann Am Thorac Soc. 2019 Jan;16(1):99-106. doi: 10.1513/AnnalsATS.201805-332OC. PMID 30417670
- [Background] Ozalevli S, Karaali HK, Ilgin D, Ucan ES. Effect of home-based pulmonary rehabilitation in patients with idiopathic pulmonary fibrosis. Multidiscip Respir Med. 2010 Feb 28;5(1):31-7. doi: 10.1186/2049-6958-5-1-31. PMID 22958625
- [Background] Rammaert B, Leroy S, Cavestri B, Wallaert B, Grosbois JM. Home-based pulmonary rehabilitation in idiopathic pulmonary fibrosis. Rev Mal Respir. 2011 Sep;28(7):e52-7. doi: 10.1016/j.rmr.2011.06.006. Epub 2011 Jul 30. PMID 21943547
- [Background] Chung BPH, Chiang WKH, Lau H, Lau TFO, Lai CWK, Sit CSY, Chan KY, Yeung CY, Lo TM, Hui E, Lee JSW. Pilot study on comparisons between the effectiveness of mobile video-guided and paper-based home exercise programs on improving exercise adherence, self-efficacy for exercise and functional outcomes of patients with stroke with 3-month follow-up: A single-blind randomized controlled trial. Hong Kong Physiother J. 2020 Jun;40(1):63-73. doi: 10.1142/S1013702520500079. Epub 2020 Feb 20. PMID 32489241
- [Background] Thorpe O, Johnston K, Kumar S. Barriers and enablers to physical activity participation in patients with COPD: a systematic review. J Cardiopulm Rehabil Prev. 2012 Nov-Dec;32(6):359-69. doi: 10.1097/HCR.0b013e318262d7df. PMID 22941449
- [Background] Stamenova V, Liang K, Yang R, Engel K, van Lieshout F, Lalingo E, Cheung A, Erwood A, Radina M, Greenwald A, Agarwal P, Sidhu A, Bhatia RS, Shaw J, Shafai R, Bhattacharyya O. Technology-Enabled Self-Management of Chronic Obstructive Pulmonary Disease With or Without Asynchronous Remote Monitoring: Randomized Controlled Trial. J Med Internet Res. 2020 Jul 30;22(7):e18598. doi: 10.2196/18598. PMID 32729843
- [Background] Borg G. Borg's perceived exertion and pain scales: Human Kinetics; 1998.
- [Background] Whitehead L. The measurement of fatigue in chronic illness: a systematic review of unidimensional and multidimensional fatigue measures. J Pain Symptom Manage. 2009 Jan;37(1):107-28. doi: 10.1016/j.jpainsymman.2007.08.019. PMID 19111779
- [Background] Reychler G, Boucard E, Peran L, Pichon R, Le Ber-Moy C, Ouksel H, Liistro G, Chambellan A, Beaumont M. One minute sit-to-stand test is an alternative to 6MWT to measure functional exercise performance in COPD patients. Clin Respir J. 2018 Mar;12(3):1247-1256. doi: 10.1111/crj.12658. Epub 2017 Jun 15. PMID 28621019
- [Background] Briand J, Behal H, Chenivesse C, Wemeau-Stervinou L, Wallaert B. The 1-minute sit-to-stand test to detect exercise-induced oxygen desaturation in patients with interstitial lung disease. Ther Adv Respir Dis. 2018 Jan-Dec;12:1753466618793028. doi: 10.1177/1753466618793028. PMID 30091679
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Chatwin M, Hawkins G, Panicchia L, Woods A, Hanak A, Lucas R, Baker E, Ramhamdany E, Mann B, Riley J, Cowie MR, Simonds AK. Randomised crossover trial of telemonitoring in chronic respiratory patients (TeleCRAFT trial). Thorax. 2016 Apr;71(4):305-11. doi: 10.1136/thoraxjnl-2015-207045. PMID 26962013
- [Background] Nolan CM, Birring SS, Maddocks M, Maher TM, Patel S, Barker RE, Jones SE, Walsh JA, Wynne SC, George PM, Man WD. King's Brief Interstitial Lung Disease questionnaire: responsiveness and minimum clinically important difference. Eur Respir J. 2019 Sep 5;54(3):1900281. doi: 10.1183/13993003.00281-2019. Print 2019 Sep. PMID 31221807